CLINICAL TRIAL: NCT04474626
Title: Single-arm Phase 2 Study of Oral Isoquercetin in Sickle Cell Disease
Brief Title: Isoquercetin in Sickle Cell Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial did not activate
Sponsor: Jeffrey Zwicker, MD (Other)
Collaborators: Quercegen Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Zwicker, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-087
Record Dates: First submitted 2020-07-06; First posted 2020-07-17 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Sickle Cell Disease; Sickle Cell-Beta0-Thalassemia
Keywords: Sickle Cell Disease; Sickle Cell-Beta0-Thalassemia; isoquercetin
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — isoquercitrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ISOQUERCETIN (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits
  - ISOQUERCETIN: Oral Study Drug, 1 time per day, per predetermined dosed per 28 treatment cycle.
  This will continue for up to 337 days.
  Interventions: Drug: Isoquercetin

INTERVENTIONS:
Drug: Isoquercetin — Oral, 1 time per day, per predetermined dosed per 28 treatment cycle.
  Other Names: IQC-950AN

SUMMARY:
This research study is being done to assess the safety and effectiveness of isoquercetin to reduce levels of soluble P-Selectin in patients with sickle cell disease. Isoquercetin is a naturally occurring flavonoid-or vitamin. You will find quercetin and isoquercetin in fruits and vegetables.

The names of the study drug involved in this study are/is:

- Isoquercetin

DETAILED DESCRIPTION:
This is a single-arm phase 2 study in adults with Sickle Cell Disease (SCD) to assess the effect of oral isoquercetin on biomarkers of endothelial and platelet activation, inflammation and ongoing blood coagulation.

* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

  * The names of the study drug involved in this study are/is: Isoquercetin
  * Participants will receive study treatment for 1 year and will be followed for 30 days after the last dose.
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.
* The U.S. Food and Drug Administration (FDA) has not approved isoquercetin as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects require an established diagnosis of sickle cell disease/homozygous hemoglobin S (SCD-SS) or sickle cell disease hemoglobin β0-thalassemia (SCD-Sβ0-thal).
* Patients on other therapy including hydroxyurea will be included.
* Age 18-50 years.
* Participants must have preserved organ and marrow function as defined below:

  * leukocytes ≥2,000/mcL
  * platelets ≥75,000/mcL
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Estimated creatinine clearance ≥45 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Subjects with no evidence of worsening over the last 4 weeks (e.g. any acute complication of SCD including but not limited to VOC, acute chest syndrome and stroke, that required unscheduled medical attention or intervention) as determined by the investigator will be included.
* Patients on anticoagulation therapy will be excluded.
* The effects of isoquercetin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of isoquercetin administration.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Please ensure exclusion criteria are clearly worded to describe participants who will not be eligible.
* Participants may not be concurrently receiving any other study agents.
* Subjects with no evidence of worsening over the last 1 month (e.g. any acute complication of SCD including but not limited to VOC, acute chest syndrome and stroke, that required unscheduled medical attention or intervention) as determined by the investigator will be included.
* Familial bleeding diathesis.
* Known diagnosis of disseminated intravascular coagulation.
* Currently receiving anticoagulant therapy.
* Currently using daily use of aspirin (>81mg daily), Clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox) (within 10 days)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to isoquercetin.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric illness/social situations that would limit study compliance.
* Pregnant women are excluded from this study because isoquercetin is a PDI inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with isoquercetin, breastfeeding should be discontinued if the mother is treated with isoquercetin. These potential risks may also apply to other agents used in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sP Selectin levels with isoquercetin | baseline to 28 Days
  Comparisons between baseline and follow-up measurements (i.e. change in sP-Selectin), will be performed using a two-tailed, paired t-test analyses.

SECONDARY OUTCOMES:
Platelet dependent thrombin generation (coagulation) | baseline to 1 year
  Laboratory values at baseline and subsequent monthly follow-up time points will be modeled using linear mixed effects regression with an autoregressive covariance structure.
sE-selectin (adhesion)-Biomarker | baseline to 1 year
  Laboratory values at baseline and subsequent monthly follow-up time points will be modeled using linear mixed effects regression with an autoregressive covariance structure.
C-reactive protein CRP | baseline to 1 year
  Laboratory values at baseline and subsequent monthly follow-up time points will be modeled using linear mixed effects regression with an autoregressive covariance structure.
Number of Participants With Treatment-Related Adverse Events | start of study treatment up to 13 months
  Sickle cell events such as SCPC, uncomplicated pain crisis, hospitalizations, emergency room visits, transfusions, acute chest syndrome and transfusion support will be summarized as annualized numbers. Statistical comparisons will be made for each patient relative to the number from the previous year using a Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu